CLINICAL TRIAL: NCT01380353
Title: Pilot Study to Test Uniformity of Transdermal Drug Delivery to the Breast Using Diclofenac Epolamine as a Model
Brief Title: Test Uniformity of Transdermal Drug Delivery to Breast Using Diclofenac Epolamine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 10B05; STU00042939 (Other: Northwestern University eIRB)
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: Women undergoing total mastectomy; Breast cancer prevention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Breast Group (Experimental): Diclofenac epolamine patch applied to the breast
  Interventions: Drug: Diclofenac epolamine patch
- Abdomen Group (Experimental): Diclofenac epolamine patch applied to the abdomen
  Interventions: Drug: Diclofenac epolamine patch

INTERVENTIONS:
Drug: Diclofenac epolamine patch — Patch (10cm X 14cm) is comprised of an adhesive material containing 1.3% diclofenac epolamine which is applied to a non-woven polyester felt backing and covered with a polypropylene film release liner [B].
  Other Names: Flecto Patch

SUMMARY:
The purpose of this study is to look for ways to improve breast cancer treatment by giving breast cancer drugs through the skin of the breast.

The drug used in this study is a diclofenac epolamine patch and is a nonsteroid anti-inflammatory pain reliever. The drug amount that gathers in the breast, after application of a patch to the skin of the breast, will be measured and compared to the amount that is found in the breast when the patch is applied to the skin of the belly.

DETAILED DESCRIPTION:
This is a randomized study where participants in group 1 will apply the diclofenac epolamine patch to the breast and participants in group 2 will apply the same drug to her abdomen. Participants are instructed to apply a new patch every 12 hours for 3 days. Total participation in this study will be for three days, ending on the day of surgery. On the day of surgery, participants will have blood drawn to measure the level of diclofenac epolamine in the body, and the final patch will be removed.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 80 years, undergoing total mastectomy for, with or without axillary surgery for diagnosis or prevention of breast cancer.
* ECOG performance status less than 2.
* Ability to understand and the willingness to sign a written informed consent.
* Participants must have normal organ and marrow function

Exclusion Criteria:

* Prior history of ipsilateral breast radiotherapy.
* Pregnant women and those who will be actively breast-feeding in the preoperative period will be excluded.
* Inability to discontinue aspirin or warfarin use during the period of participation.
* Known allergy to diclofenac epolamine, or aspirin, diclofenac (Cataflam, Voltaren), or another non-steroidal anti-inflammatory drug (NSAID).
* Renal failure

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11-12 (Actual); Study Completion 2012-11-12 (Actual)

PRIMARY OUTCOMES:
Compare concentrations of diclofenac epolamine patch when applied to breast vs. abdomen | after 3 days of treatment prior to surgery
  The primary objective of this protocol will demonstrate that diclofenac epolamine patch applied to the skin of the breast for three days (1, 2) prior to surgery will result in significantly higher drug concentrations in the breast than the same dose applied to the abdominal skin for the same duration of time.

SECONDARY OUTCOMES:
Determine how the concentrations of the study patch is distributed in the breast. | after three days of treatment prior to surgery
  To establish that the diclofenac epolamine drug concentrations achieved in the breast have no significant fall-off with increasing distance from the site of application. Therefore, uniform therapeutic concentrations are achieved throughout the breast with a single site of local transdermal therapy (LTT).

CONTACTS AND LOCATIONS:
Overall Officials: Seema Khan, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States